CLINICAL TRIAL: NCT01833234
Title: Questionnaire Development for a Comprehensive Scale to Measure the Impact of Epilepsy on Life.
Brief Title: Epilepsy Impact Scale
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: James & Carrie Anderson Fund for Research in Epilepsy (Unknown)
Responsible Party: Principal Investigator, Robert S. Fisher, M.D., Ph.D., Professor of Neurology, Stanford University
Other Study IDs: Stanford Epilepsy IRB 20523
Record Dates: First submitted 2013-03-29; First posted 2013-04-16 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Epilepsy
Keywords: epilepsy; quality of life; seizure severity; antiepileptic drug side effects; questionnaire; patient reported outcomes
MeSH Terms: conditions — Epilepsy | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- People with epilepsy: People with epilepsy who have have had at least one seizure in the prior year.
  Interventions: Other: Interviews and questionnaires

INTERVENTIONS:
Other: Interviews and questionnaires

SUMMARY:
The investigators are developing a questionnaire that can quickly measure the impact that epilepsy has on a person's life. This questionnaire will be useful in following whether the impact of epilepsy increases, decreases or stays the same over time. The results also may point out areas that would benefit from discussion or attention in visits with your doctor.

DETAILED DESCRIPTION:
The investigators have used a set of broad open-ended questions about the impact of epilepsy on a person's life to formulate a long list of questions to characterize the impact the seizures, medications, and comorbidities that you are having. In the future, this will be boiled down to a short list of questions.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more.
2. Patient has had at least 1 seizure in the past 365 days.
3. Patient can speak and understand English.

Exclusion Criteria:

1. Patients suspected of having one of the imitators of epilepsy, for example, syncope, sleep disorder, psychogenic nonepileptic seizures, will be excluded, even if they also have epileptic seizures.
2. Patients unwilling to spend the time doing the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the Stanford Epilepsy Center who have had a seizure in the past year and agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Validation of a concise question set | Up to 1 year for question set validation, data presentation within up to 1.5 years

SECONDARY OUTCOMES:
Correlation of subscales | Up to 1.5 years
  Correlation of subscales of the study questionnaire with previously validated scales, including QoLiE-39, NHS Seizure Severity Scale, Liverpool side effects scale, Beck Depression Index

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Fisher, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States